CLINICAL TRIAL: NCT00776646
Title: An Open Label, Balanced, Randomized, Two-Treatment, Two-Period, Two- Sequence, Single-Dose, Crossover Bioavailability Study Comparing Hydrochlorothiazide 50 mg Tablet of Ohm Laboratories (A Subsidiary of Ranbaxy Pharmaceuticals USA) With Hydrochlorothiazide 50 mg Tablet of IVAX Pharmaceuticals in Healthy, Adult, Human, Male Subjects Under Fasting Condition
Brief Title: Bioequivalence Study of Hydrochlorothiazide 50mg Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Collaborators: IPCA Laboratories Ltd. (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 107_HYDRO¬_06
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: bioequivalence hydrochlorothiazide 50 mg tablet fasting conditions
MeSH Terms: interventions — Hydrochlorothiazide; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): hydrochlorothiazide 50 mg tablet
  Interventions: Drug: hydrochlorothiazide 50 mg tablet
- 2 (Active Comparator): hydrochlorothiazide 50 mg tablet
  Interventions: Drug: hydrochlorothiazide 50 mg tablet

INTERVENTIONS:
Drug: hydrochlorothiazide 50 mg tablet

SUMMARY:
To compare the single-dose oral bioavailability of hydrochlorothiazide 50 mg tablet of Ohm Laboratories (A subsidiary of Ranbaxy pharmaceuticals USA) with hydrochlorothiazide 50 mg tablet of IVAX Pharmaceuticals, USA in healthy, adult, human, male subjects under fasting condition

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomised, two-treatment, two-period, two- sequence, single-dose, crossover bioavailability study comparing hydrochlorothiazide 50 mg tablet, containing 50 mg of hydrochlorothiazide of Ohm Laboratories (A subsidiary of Ranbaxy pharmaceuticals USA) with hydrochlorothiazide 50 mg tablet, containing 50 mg of hydrochlorothiazide of IVAX Pharmaceuticals, in healthy, adult, human, male subjects under fasting condition.

During the course of the study safety parameters assessed were vital signs, clinical examination, medical history and clinical laboratory safety tests (hematology, biochemical, serology parameters and urine analysis) at base line. Laboratory parameters of hematology and biochemistry were repeated at the end of the study. In addition serum electrolytes Sodium, Potassium and Chloride were measured on admission and at the discharge of each period.

A total of 36 subjects were randomized to receive single oral dose of hydrochlorothiazide 50 mg tablet and 31 subjects completed both the periods of the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45 years.
* Were neither overweight nor underweight for his height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
* Had voluntarily given written informed consent to participate in this study.
* Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.

Exclusion Criteria:

* - Had history of allergy or hypersensitivity to hydrochlorothiazide or any other sulphonamide derived drugs.
* Had history of diarrhoea, vomiting or headache within past two weeks
* Had history of hypotension (systolic BP<100 mmHg)
* Had history of allergy or bronchial asthma
* Had history of muscle cramps or muscle weakness
* Had history of any anaphylactic reactions, necrotizing angiitis (vasculitis and cutaneous vasculitis), respiratory distress including pneumonitis and pulmonary edema, photosensitivity, fever, urticaria, rash, purpura, Systemic Lupus Erythematoses(SLE)
* Had history of aplastic anemia, agranulocytosis, leukopenia, hemolytic anemia, thrombocytopenia
* Had history of anuria or history/evidence of any renal disorder including renal failure, renal dysfunction, interstitial nephritis.
* Had history of erythema multiforme including Stevens- Johnson syndrome or exfoliative dermatitis including toxic epidermal necrolysis
* Had history of pancreatitis
* Had history/evidence of jaundice or any hepatic or gall bladder disease
* Had history of hyperglycemia, glycosuria, hyperuricemia or gout.
* The subject had a history/evidence of any electrolyte imbalance, serum sodium < 135 mEq/L, serum potassium < 3.5 mEq/ L.
* Had any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
* Had presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
* Had presence of values, which are significantly different from normal, reference and/or judged clinically significant for haemoglobin, total white blood cells count, differential WBC count or platelet count.
* Had positive for urinary screen testing of drugs of abuse (opiates or cannabinoids)
* Had presence of values, which are significantly different from normal, reference ranges and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
* Had clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), epithelial cells (>4/HPF), glucose (positive) or protein (positive).
* Had clinically abnormal ECG or Chest X-ray.
* Had history of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes or glaucoma.
* Had history of any psychiatric illness, which may impair the ability to provide, written informed consent.
* Were regular smokers who smoke more than 10 cigarettes daily or have difficulty abstaining from smoking for the duration of each study period.
* Had history of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or have difficulty in abstaining for the duration of each study period.
* Had used any enzyme modifying drugs within 30 days prior to Day 1 of this study.
* Had participated in any clinical trial within 12 weeks preceding Day 1 of this study.
* Subjects who, through completion of this study, would have donated and/or lost more than 350 mL of blood in the past 3 months.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-05; Primary Completion 2006-06 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html